CLINICAL TRIAL: NCT01758211
Title: Blood Oxygen Level Dependent fMRI Navigation for Function Protection in Intracranial Arteriovenous Malformation Surgery: a Multicenter Prospective Randomized Controlled Single Blind Clinical Trial
Brief Title: Functional Magnetic Resonance Imagine(fMRI)Navigation in Intracranial Arteriovenous Malformation Surgery
Acronym: FMRINAVMS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, MD, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVM-125-FMRI
Record Dates: First submitted 2012-12-26; First posted 2013-01-01 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Intracranial Arteriovenous Malformations
Keywords: Intracranial Arteriovenous Malformations; Functional Magnetic Resonance Imaging; Neuronavigation
MeSH Terms: conditions — Intracranial Arteriovenous Malformations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fMRI guided resection of AVM (Experimental): fMRI Navigation AVM resection in AVM patients
  Interventions: Procedure: fMRI Navigation AVM resection
- conventional AVM resection (Active Comparator): conventional resection of AVM
  Interventions: Procedure: conventional resection

INTERVENTIONS:
Procedure: fMRI Navigation AVM resection — intraoperative fMRI navigation guided resection in AVM patients
  Arms: fMRI guided resection of AVM
Procedure: conventional resection — conventional resection in AVM patients
  Arms: conventional AVM resection

SUMMARY:
Little is known about the effect of fMRI navigation in the intracranial arteriovenous malformation surgery. The investigators aim to perform a multicenter prospective randomized single -blind clinical trial to assess the effect and safety of fMRI navigation in the brain arteriovenous malformation surgery.

DETAILED DESCRIPTION:
Intracranial arteriovenous malformations (AVMs) are congenital lesions that consist of multiple arteries and veins, connecting as a fistula without an intervening normal capillary bed. Surgical removal is thought as a major treatment option for AVMs. However, compared with stereotaxic radiosurgery and endovascular embolization, microsurgery of AVMs is regarded with high mortality and morbidity, particular for high level classification AVMs .

Blood oxygen level dependent fMRI can be used to mapping the motor and language regions of the brain noninvasively. It has been one of the most advanced functional imaging techniques and it has quickly grown to be a vital tool for clinical and cognitive neuroscience research. Many clinical researches have been reported about the utility of fMRI in brain tumor surgery. However, the effect of fMRI navigation for neurofunction protection in the intracranial arteriovenous malformation surgery was unclear.

We aim to perform a multicenter prospective randomized single -blind clinical trial to assess the safety and effect of fMRI navigation in the intracranial AVMs surgery. We hypothesize that application of blood oxygen level dependent fMRI is able to improve long term prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of intracranial AVM by DSA/CT/MRI
2. Age from 12-60 years
3. Be suitable for microsurgery treatment
4. All patients are able to cooperate with the fMRI examination
5. All patients gave written informed consent

Exclusion Criteria:

1. Patients with age < 12 years or > 60 years
2. Various conditions unable to meet the indications for microsurgery treatment
3. Intracranial hemorrhage need emergency surgery
4. Patients can not cooperate with fMRI examination

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
modified Ranking Scale | six months after operation
  The scale runs from 0-6, running from perfect health without symptoms to death. 0-No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead.

SECONDARY OUTCOMES:
Postoperative complications | six months after operation
  Post operative epilepsy seizure, hemorrhage,infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, MD, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li M, Jiang P, Guo R, Liu Q, Yang S, Wu J, Cao Y, Wang S. A Tractography-Based Grading Scale of Brain Arteriovenous Malformations Close to the Corticospinal Tract to Predict Motor Outcome After Surgery. Front Neurol. 2019 Jul 17;10:761. doi: 10.3389/fneur.2019.00761. eCollection 2019. PMID 31379715
- [Derived] Li D, Jiao YM, Wang L, Lin FX, Wu J, Tong XZ, Wang S, Cao Y. Surgical outcome of motor deficits and neurological status in brainstem cavernous malformations based on preoperative diffusion tensor imaging: a prospective randomized clinical trial. J Neurosurg. 2019 Jan 1;130(1):286-301. doi: 10.3171/2017.8.JNS17854. Epub 2018 Mar 16. PMID 29547081
- [Derived] Lin F, Jiao Y, Wu J, Zhao B, Tong X, Jin Z, Cao Y, Wang S. Effect of functional MRI-guided navigation on surgical outcomes: a prospective controlled trial in patients with arteriovenous malformations. J Neurosurg. 2017 Jun;126(6):1863-1872. doi: 10.3171/2016.4.JNS1616. Epub 2016 Jul 1. PMID 27367242
- [Derived] Zhao B, Cao Y, Zhao Y, Wu J, Wang S. Functional MRI-guided microsurgery of intracranial arteriovenous malformations: study protocol for a randomised controlled trial. BMJ Open. 2014 Oct 23;4(10):e006618. doi: 10.1136/bmjopen-2014-006618. PMID 25341453